CLINICAL TRIAL: NCT03469154
Title: Sustainable Solutions for Paediatric Basic Life Support Training in Day Care Centres: A Comparative Effectiveness Trial
Brief Title: Sustainable Solutions for Paediatric Basic Life Support Training in Day Care Centres
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Asbjørn Hasselager,MD, Principal investigator, Copenhagen Academy for Medical Education and Simulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1
Record Dates: First submitted 2018-02-22; First posted 2018-03-19 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Cardiopulmonary Resuscitation; Education; Medical Emergencies
Keywords: Layperson; Paediatric Basic life Support; education

STUDY DESIGN:
Intervention Model Description: Two parallel groups. Participants randomised to either dyad training or instructor led training.
  Dyad training in pairs guided by instructional videos Instructor led training with maximum 6 participants per instructor.
Who Masked: Outcomes Assessor
Masking Description: After training participants demonstrate skills in a standardised scenario test with children resuscitation manikins. All tests are video recorded. Participants in videos identified by a unique id number. Training method is not mentioned in videos. Assessors have no knowledge on the relation between group and unique id (are blinded for the interventions). Assessors assess videos of all participants in a randomised order .
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dyad training (Experimental): The participants in this arm will train in teams of two. Participants will be instructed in paediatric basic life support by instructional videos in a computer programme and train on children resuscitation manikins. Training involves recognition of cardiac arrest, cardio-pulmonary resuscitation and foreign body airway obstruction management. The training involves series of short video clips and following exercises. Each participant performs the exercise and the other gives feedback. Afterwards roles are changed. The procedure is done for all exercises after a video clip. The duration of the training is maximum 50 minutes
  Interventions: Other: Dyad training method
- Instructor led training (Active Comparator): Participants train in courses of up to 6 participants with an instructor. Training content is identical to dyad training content involving: recognition of cardiac arrest, cardio-pulmonary resuscitation and foreign body airway obstruction management.
  Skills are instructed by an instructor using af 4 step approach (1. show skills, 2. show with explanation, 3. participants instruct instructor, 4. participants performs the skills on resuscitation manikins). Training is maximum two hours but course duration is adjusted to number of participants two allow for similar hands-on time per participant as in the experimental arm.
  Interventions: Other: Instructor led training method

INTERVENTIONS:
Other: Dyad training method — The training model for paediatric basic life support for laypersons involves a course based on pairs training together guided by instructional videos and with hands-on practice on resuscitation manikins.
  Arms: Dyad training
Other: Instructor led training method — The training model for paediatric basic life support for laypersons involves a course led by an instructor including hands-on practice on resuscitation manikins.
  Arms: Instructor led training

SUMMARY:
In a randomised non-inferiority trial the investigators examine two training interventions to train paediatric basic life support to laypersons: Dyad training vs Instructor led training.

For dyad training two participants are guided by video instructions and perform exercises on children resuscitation manikins. The participants take turn to complete the exercises and provide feedback to their peer. The duration is up to 50 minutes Instructor led training of paediatric basic life support in instructor led courses with up to 6 participants per course with hands-on training on children resuscitation manikin. The duration of the courses is up to two hours.

Instructor led training represents the common gold standard for training Paediatric Basic Life Support, however it is inflexible and uses a lot of resources. Dyad training provides a low cost solution with improved flexibility. Consequently a non-inferiority design is chosen as the benefits of dyad training with the same learning outcomes favours the dyad training method.

Prior to the training both groups are informed about and have access to a website with videos, quizzes, pictures and text information on paediatric basic life support and foreign body airway obstruction management.

DETAILED DESCRIPTION:
Introduction Paediatric Basic Life support (PBLS) training is essential for acquisition of resuscitation skills. Trained laypersons are more likely to provide bystander cardiopulmonary resuscitation. The skills are important if life-threatening incidents occur as immediate bystander response is needed to improve survival and neurological outcomes for critically ill children. Previously most training has been conducted by instructor-led training courses of small groups. The courses are fairly good at learning the skills, but the skills acquired still deteriorate in a period as quickly as six months. To increase survival of children there is a need for teaching PBLS skills to large communities. Instructor-led training is not suitable for this task due to the need of very large numbers of instructors, the short retention spans, the inflexibility of the course planning and the economic costs of having small groups training with an expensive instructor thus emphasising needs for alternative training strategies.

Alternative approaches to community based learning of PBLS have not been examined in larger scales and especially not in the lights of feasibility, retention and costs. Improving retention of skills or developing feasible quick retraining methods with relevant intervals for the purpose of maintaining PBLS skills remains a challenge.

This study examines these problems by conducting a study of an alternative approach to PBLS training for the community of employees in day care centres using dyad training. If successful, the training method could provide flexible training, improve retention, reduce costs and be suitable for training large communities.

Dyad training In the Dyad training method learners work together in pairs to acquire skills. The participants take turns in performing the practical skills and the other observes and gives feedback. In other medical settings dyad training has been found effective in skills training especially for novices and in short courses. The dyad training studies have been limited to small numbers of health care professional participants in simulated settings. Possible explanations of these effects include observational processing, psychomotor, cognitive and social factors and the mirror neuron system. The use of dyad partners allows learners to observe, support and feedback each other during practice and thereby reduce cognitive load and support cognitive co-construction. The active role as dyad observer has been suggested to let participants set higher goals for own performance, increase motivation by inducing a competitive component and increase responsibility for training which in all cases may enhance the cognitive processing and increase learning. The learning strategy has not been studied for workplace-based skills learning, in PBLS nor for larger groups of lay persons. Dyad training in this study is assisted and facilitated by computer based video instruction as other studies have found it to be effective for novice training. Consequently the presented learning method does not involve an instructor and presents an alternative to traditional skills training which could prove efficient, feasible, flexible and reduce costs. Secondly the training method has a potential for easy up scaling to larger groups/communities. Some studies have found positive correlations between simulation assessment and patient-related outcomes, linking the PBLS training to real life incidents.

The aim of this study is in a randomised control trial to examine if dyad training and E-learning (dyads guided by computer programme videos) as a learning model is non-inferior to instructor led training regarding acquisition of PBLS practical skills and self-efficacy in lay persons. The investigators want to examine if the dyad training positive effects described in literature can be applied to short training courses in a broader population. Second the investigators want to examine if the learning and retention of PBLS skills is affected by the training methods.

Prior to the training both groups have access to a website with videos, quizzes, pictures and text information on paediatric basic life support and foreign body airway obstruction management.

The investigators hypothesise that dyad training and E learning is non-inferior or equivalent compared to instructor led practical skills training. The hypothesis emerges from data obtained in focus group interviews stating that employees are used to work in teams, find PBLS training very important, want to engage in this form of training and lack PBLS competencies. Incidents in day care centres are handled in teams hence dyad training is similar to real life situations in day care centres and this may increase motivation and learning. If incidents requiring PBLS are to be performed in day care centres it will be in a stressful environment with reduced individual cognitive capacities thus supporting teamwork and sharing resources. This may be strengthened by the dyad training method.

Real transfer studies cannot be performed regarding PBLS but training close to realities (i.e. in groups of well-known colleagues) may facilitate easier transfer to real incidents.

Interviews have indicated that instructor-led training might boost immediate self-confidence and potentially the performance right after a course but may deteriorate fast when course and instructor support stops. It is hypothesized that the possible enhanced cognitive processing after the course suggested in dyad training may improve performance and retention of skills after the course compared to individual instructor-led training.

In addition to the analysis mentioned above elf-efficacy on acquired skills in PBLS will be examined in questionnaires as it is important for bystanders' willingness to act.

The assessment tool to assess video recorded scenario tests has been examined for validity evidence winter 2017/2018. Consequently blinded assessors are rating the videos in January through March 2018 and no analysis of the results has taken place before the clinicaltrials.gov registration.

ELIGIBILITY:
Inclusion Criteria:

* Working with children under seven years of age for >20 hours/week
* Physically able to participate in tests

Exclusion Criteria:

* Any basic life support training within 1 year from training day
* Trained health professional

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
Paediatric basic life support skill level immediately after training | Participant performs the tests of approximately 3-5 minutes, up to one hour after the course finalization.
  All participants participate in video recorded standardised scenario tests on resuscitation manikins just after the training course for paediatric basic life support. The videos are rated by blinded assessors using a developed assessment tool for laypersons paediatric basic life support (validity evidence study currently under preparation for publication) - The assessment tool is based on internationally identified assessment items from a delphi consensus study (see references).
Foreign body airway obstruction management skill level immediately after training | Participant performs the tests of approximately 3-5 minutes up to one hour after the course finalization.
  All participants participate in video recorded standardised scenario tests on resuscitation manikins just after the training course for foreign body airway obstruction management. The videos are rated by blinded assessors using a developed assessment tool for laypersons paediatric basic life support (validity evidence study currently under preparation for publication) - The assessment tool is based on internationally identified assessment items from a delphi consensus study (see references).

SECONDARY OUTCOMES:
Retention test of paediatric basic life support skills assessed by standardised scenario tests | 14 days after training
  By randomisation one third of the participants in the primary outcome 1 measure participate in a test similar to the primary outcome measure 1.
Retention test of paediatric basic life support skills assessed by standardised scenario tests | 1 month after training
  By randomisation one third of the participants in the primary outcome measure 1 participate in a test similar to the primary outcome measure 1.
Retention test of paediatric basic life support skills assessed by standardised scenario tests | 3 months after training
  By randomisation one third of the participants in the primary outcome measure 1 participate in a test similar to the primary outcome measure 1.
Retention test of foreign body airway obstruction management skills assessed by standardised scenario tests | 14 days after training
  The secondary outcome 1 participants participate in a test similar to the primary outcome measure (outcome 2).
Retention test of foreign body airway obstruction management skills assessed by standardised scenario tests | 1 month after training
  The secondary outcome 2 participants participate in a test similar to the primary outcome measure (outcome 2).
Retention test of foreign body airway obstruction management skills assessed by standardised scenario tests | 3 months after training
  The secondary outcome 3 participants participate in a test similar to the primary outcome measure (outcome 2).
Self-efficacy by questionaires | Up to 10 minutes after training
  All participants examined for self-efficacy on foreign body airway obstruction and paediatric basic life support skills. Immediately after the training course.
Self-efficacy by questionaires | 14 days after training
  Secondary outcome 1 participants examined by questionaires on self-efficacy on foreign body airway obstruction and paediatric basic life support skills. Immediately before the retention tests.
Self-efficacy by questionaires | 1 month after training
  Secondary outcome 2 participants examined by questionaires on self-efficacy on foreign body airway obstruction and paediatric basic life support skills. Immediately before the retention tests.
Self-efficacy by questionaires | 3 months after training
  Secondary outcome 3 participants examined by questionaires on self-efficacy on foreign body airway obstruction and paediatric basic life support skills. Immediately before the retention tests.

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn Hasselager, MD, Principal Investigator — Copenhagen Academy for Medical Education and Simulation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hasselager AB, Lauritsen T, Kristensen T, Bohnstedt C, Sonderskov C, Ostergaard D, Tolsgaard MG. What should be included in the assessment of laypersons' paediatric basic life support skills? Results from a Delphi consensus study. Scand J Trauma Resusc Emerg Med. 2018 Jan 18;26(1):9. doi: 10.1186/s13049-018-0474-5. PMID 29347956